CLINICAL TRIAL: NCT03149263
Title: Evaluation of the Effect of the Presence Of Clowns on Pain and Anxiety Seen During Injections Botulinum Toxin in Child
Acronym: CLOWN-TOX
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CLOWN-TOX
Record Dates: First submitted 2016-08-12; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Cerebral Palsy; Muscle Hypertonia
Keywords: botulinum toxin; anxiety reduction; pain reduction; medical clowns; distraction
MeSH Terms: conditions — Cerebral Palsy; Muscle Hypertonia | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Toxin-clown: Botulinum toxin injections are carried out according to the usual injection protocol.
  40 children will be included into the arm toxin with clown distraction. During injections, clowns take information with the doctor before the procedure on the child's pathology, the cognitive level, the number of injections. During injections, clowns fit and distraction can change depending on the reaction of the child to their intervention.
  Interventions: Behavioral: distraction
- Toxin-usual distraction: 40 children will be included into the arm "toxin with usual distraction" The usual distraction involves discussion with the child, and its accompanying its interests, to define the use of music, songs, television, video games or other distraction during the session. If the first distraction doesn't work, it's possible to switch to another distraction during injections
  Interventions: Behavioral: distraction

INTERVENTIONS:
Behavioral: distraction — Children will all benefit toxin injections with the same protocol. Only the distraction will be different during the session: either the children will have a distraction realized by the team of clowns / or children will benefit a classic distraction (TV, music, ...)

SUMMARY:
In children requiring botulinum toxin injections, improving supervisory procedures of injection sessions to reduce pain and improve the experience of this invasive procedure is needed. The intervention of medical clowns seems very interesting in this goal, but its effectiveness has not been proven within the botulinum toxin injections. The objective of the study is to evaluate in terms of profit the presence or absence of clowns during a session of botulinum toxins by determining their impact on pain and anxiety felt among children and their carers

DETAILED DESCRIPTION:
In the literature, the presence of clowns allows a major reduction of pain and anxiety in children and their accompanying in various medical and hospital surgical settings. A previous study on a population of 60 children was conducted to assess the impact of the presence of clowns during the production of botulinum toxin injection in children but not confirming the benefit of their participation in carrying this medical procedure. The results of this study are opposed to current scientific data. Their impact clown assessment criteria seem however insufficient to actually support the conclusion as to the ineffectiveness of distractibility clowns in this specific medical procedure iterative injection of botulinum toxin.

The objective of the study is to evaluate the pain and anxiety before and after the botulinum toxin injection session in children and hetero-assessment of pain and anxiety by accompanying depending on the presence or not of clown. The second objectives are the evaluation of the course of the session by the injector doctor, the accompanying of the child and to evaluated the effect of distraction during the toxin of the clown or the usual distraction (music, movie...)

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 18 years
* Children with a neurogenic spasticity (cerebral palsy, spastic paraplegia, head trauma ...)
* Children with muscular pains orthopedic disorders (POPB, equino varus, ..)
* Botulinum Toxin Injection functional target, improvement in pain or amplitudes
* First injection or repeated injections of toxins
* No opposition formalized

Exclusion Criteria:

* Children between 0 and 1 year
* Opposition formalized to the data use

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children receiving botulinum toxin in local pediatric day hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Pain assessment by a hetero evaluator at the time of toxin injections | 1 hour
  Evaluation of the pain child during botulinum toxin with the FLACC (Face Legs Activity Cry Consolability) by a hetero evaluator

SECONDARY OUTCOMES:
Evaluation of anxiety before the injections of botulinum toxins by the child and assessment by a accompanying person | 1 hour
  evaluation of the anxiety before the botulinum toxin by the use of a VAS anxiety scale for the children and their accompanying person
Evaluation of pain and anxiety after the botulinum toxin injection session in children and the accompanying person depending on the presence or not of clowns | 1 hour
  evaluation of the anxiety after the botulinum toxin by the use of a VAS anxiety scale for the children and their accompanying person
Evaluation of the course of the session of botulinum toxin by the injector doctor | 1 hour
  Evaluation of the progress of the botulinum toxins session by the injector doctor on a scale of 0-4 (0 bad conduct and 4 very smooth conduct of the session)
Evaluation of the course of the session of botulinum toxin by the accompanying person | 1 hour
  Evaluation of the progress of the botulinum toxins session by the accompanying person on a scale of 0-4 (0 bad conduct and 4 very smooth conduct of the session)
Evaluation of the effect of distraction during the session of botulinum toxin with the usual distraction (music, movie, ...) or the participation of the clown(s) distraction | 1 hour
  Evaluation of the effect of distraction establishment on a scale of 0 to 4 estimated in the accompanying person (0 bad conduct and 4 very smooth conduct of the session)

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Houx, MD, Principal Investigator — Physical Medical and Rehabilitation, CHRU Brest, France
Locations (1):
- Houx, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vagnoli L, Caprilli S, Robiglio A, Messeri A. Clown doctors as a treatment for preoperative anxiety in children: a randomized, prospective study. Pediatrics. 2005 Oct;116(4):e563-7. doi: 10.1542/peds.2005-0466. PMID 16199685
- [Background] Hansen LK, Kibaek M, Martinussen T, Kragh L, Hejl M. Effect of a clown's presence at botulinum toxin injections in children: a randomized, prospective study. J Pain Res. 2011;4:297-300. doi: 10.2147/JPR.S23199. Epub 2011 Sep 21. PMID 22003302
- [Result] Molenaers G, Schorkhuber V, Fagard K, Van Campenhout A, De Cat J, Pauwels P, Ortibus E, De Cock P, Desloovere K. Long-term use of botulinum toxin type A in children with cerebral palsy: treatment consistency. Eur J Paediatr Neurol. 2009 Sep;13(5):421-9. doi: 10.1016/j.ejpn.2008.07.008. Epub 2008 Nov 1. PMID 18977158
- [Result] Schroeder AS, Berweck S, Lee SH, Heinen F. Botulinum toxin treatment of children with cerebral palsy - a short review of different injection techniques. Neurotox Res. 2006 Apr;9(2-3):189-96. doi: 10.1007/BF03033938. PMID 16785117
- [Result] Brochard S, Blajan V, Lempereur M, Le Moine P, Peudenier S, Lefranc J, Remy-Neris O. Effectiveness of nitrous oxide and analgesic cream (lidocaine and prilocaine) for prevention of pain during intramuscular botulinum toxin injections in children. Ann Phys Rehabil Med. 2009 Dec;52(10):704-16. doi: 10.1016/j.rehab.2009.09.001. Epub 2009 Oct 6. PMID 19854692
- [Result] Bayon-Mottu M, Gambart G, Deries X, Tessiot C, Richard I, Dinomais M. Pain during injections of botulinum toxin in children: Influence of the localization technique. Ann Phys Rehabil Med. 2014 Dec;57(9-10):578-86. doi: 10.1016/j.rehab.2014.09.010. Epub 2014 Oct 8. PMID 25454692
- [Derived] Houx L, Dubois A, Brochard S, Pons C. Do clowns attenuate pain and anxiety undergoing botulinum toxin injections in children? Ann Phys Rehabil Med. 2020 Oct;63(5):393-399. doi: 10.1016/j.rehab.2018.12.004. Epub 2019 Jan 29. PMID 30708069